CLINICAL TRIAL: NCT06397664
Title: A Quantitative and Qualitative Study on the Impact of Chronic Adolescent Skin Conditions on Sexual Health
Brief Title: The Impact of Chronic Adolescent Skin Conditions on Sexual Health
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Tess Mcpherson, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 329926
Record Dates: First submitted 2024-04-24; First posted 2024-05-03 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Psychological; Sexual Dysfunction; Adolescent Development; Interaction, Social; Dermatologic Disease
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Skin Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Background: Skin conditions are common in young people and are known to adversely affect emotional well-being and quality of life in a range of ways, including negative impact on intimate relationships. However, despite its importance, it has been shown that dermatology consultations rarely address issues like genital skin involvement or sexual dysfunction. Furthermore, there is currently very little data on the scale of the problem, risk factors, psychological impact of skin on sexual function or understanding of the most appropriate ways to manage it in this age group.

Research aims: The Dermatology department at Oxford University Hospitals National Health Service Trust (Oxford, United Kingdom) have already set up an award-winning specialist dermatology service for young people with embedded psychological support. This study further explores how services can be improved by evaluating the impact of chronic skin conditions on quality of life and sexual dysfunction in adolescents. By identifying the associated risk factors, recommendations can be made to effectively meet the physical and mental health needs of adolescents.

Design and methods: The study will gain perspectives from follow-up patients aged 17 - 25 years seen by the Dermatology departments in Oxford University Hospitals National Health Service Trust (Oxford, United Kingdom). They will complete an online anonymous survey to share how their skin condition affects their quality of life, including sex and intimacy, and how services can be improved to meet their needs. In-depth interviews will then be conducted in those who volunteer, to better understand the nuances of unmet needs. Participation is voluntary.

Dissemination: Results of the research will be disseminated by national and international conferences, publications in academic dermatology journals and collaborations with other NHS departments. Improvements will be made to the local adolescent dermatology service as a result and shared via local meetings and posters.

ELIGIBILITY:
Inclusion Criteria:

* The participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 17-25 (inclusive).
* Diagnosed with a long-term skin condition and seen as a follow-up patient in the clinic.
* Recruited from Paediatric/Adolescent, General and Acne clinics under the Oxford University Hospitals National Health Service Trust Dermatology Department.
* Fluent in English (reading and writing).

Exclusion Criteria:

* No informed consent was given to participate in the study or use the data for research purposes.
* No capacity to make an informed decision to consent.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants are adolescents aged 17-25 (inclusive) who have a chronic skin condition and are seen as follow-up patients under the Oxford University Hospitals National Health Service Trust Dermatology Department.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Scores from the modified T-QOL (Teenager's Quality of Life Index) to 1 year | Baseline (Retrospective study)
  T-QOL is modified to 1 year to reflect the impact of chronic skin conditions. Scores range from 0 (least impairment on quality of life) to 36 (greatest impairment on quality of life).
  It is self-reported and validated.
Scores from the IIEF (International Index of Erectile Function) | Baseline (Retrospective study)
  IIEF reflects 5 domains - male erectile function (maximum score 30) and intercourse satisfaction (maximum score 15), orgasmic function, sexual desire, intercourse satisfaction, overall satisfaction (maximum scores of 10). Low scores correlate with worse outcomes.
  It is self-reported and validated.
Scores from the FSFI (Female Sexual Function Index) | Baseline (Retrospective study)
  FSFI reflects 6 domains - female sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. All domains have a maximum score of 6 and can be totalled. Low scores correlate with worse outcomes.
  It is self-reported and validated.
Scores from the PHQ-9 (Patient Health Questionnaire) | Baseline (Retrospective study)
  PHQ-9 is a diagnostic tool to monitor depression severity. Scores range from 0 (no depression) to 27 (severe depression).
  It is self-reported and validated.
Scores from the GAD-2 (Generalised Anxiety Disorder 2-item) | Baseline (Retrospective study)
  GAD-2 initially screens for generalised anxiety disorder. The scores range from 0 (unlikely to have GAD) to 6 (most likely to have GAD).
  It is self-reported and validated.

SECONDARY OUTCOMES:
A narrative synthesis detailing risk factors impacting sexual function in adolescents with chronic skin conditions | Baseline (Retrospective study)
  A narrative synthesis derived from the thematic analysis of at least 20 in-depth semi-structured interviews, using a constant comparison and mind-mapped approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Churchill Hospital, Oxford University Hospitals NHS Trust, Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No